CLINICAL TRIAL: NCT03303898
Title: ASYMPTOMATIC CARRIER OF LEISHMANIA INFANTUM, MEDISERRANEAN VISCERAL LEISHMANIOSIS AGENT: STUDY OF IMMUNE RESPONSE - POSTULATE PRIOR TO HUMAN VACCINAL TRIALS Immune Response of Asymptomatic Carriers to L. Infantum
Brief Title: ASYMPTOMATIC CARRIER OF LEISHMANIA INFANTUM, MEDISERRANEAN VISCERAL LEISHMANIOSIS AGENT: STUDY OF IMMUNE RESPONSE -
Acronym: Asymptoleish
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-AOI-04
Record Dates: First submitted 2017-10-03; First posted 2017-10-06 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Leishmaniasis, Cutaneous
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- asymptomatic carriers (Other)
  Interventions: Procedure: Blood sampling
- uninfected patient (Other)
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — sampling of 7 blood tubes

SUMMARY:
Leishmaniasis is considered by the WHO as emerging and uncontrolled diseases. They are the second leading cause of death and the fourth leading cause of morbidity in tropical diseases. Leishmaniasis is parasitic reticulo-endotheliosis, the pathogenic agent of which is a flagellated protozoan belonging to the genus Leishmania. It is estimated that there are about 2 million new cases per year. Effective treatments against visceral leishmaniasis are few and resistance problems appear. To date, only a canine vaccine is available protecting dogs from the development of canine leishmaniasis to L. infantum. In man, in parallel clinical cases, leishmaniasis is characterized by a large number of asymptomatic carriers. This is the case in the Alpes-Maritimes where 50% of the inhabitants of the hinterland of Nice are carriers of the parasite.

the investigators wish to study the protective immune response to the parasite and more particularly to the asymptomatic carriers. Indeed, these patients were infected with the parasite and did not develop the disease. Understanding the protective immune response in these patients against the parasite is therefore paramount in the development of a human leishmaniasis vaccine.

For this purpose, the investigator wants to make an ex vivo study of the immune response of lymphocytes coming from asymptomatic carriers after stimulation by Leishmania vaccine peptides. It also wants to describe the immune response, after stimulation by these peptides, in the lymphocytes of subjects asymptomatic carriers and lymphocytes from subjects not infected with the parasite and comparing them. This study is unicentric and non-randomized. It wishes to recruit 20 asymptomatic carriers of L. Infantum and 10 uninfected subjects. They will be selected from our database. A simple blood sample will be taken. After verification by quantitative PCR and western blotting of their status towards leishmaniasis, the team will divide them into two groups (asymptomatic or healthy). Then the blood samples will be sent to the team of Jean Loup Lemesre of the Laboratory INTERTRYP - UMR177 of the IRD in Montpellier. ELISPOT analysis and assay of cytokines and proteases to describe the immune response of the two groups and to compare them. In addition, cell typing will be performed by flow cytometry to determine the type of lymphocytes involved in the immune response against Leishmania peptides. HLA typing will also be performed to validate the HLA coverage of the peptides tested. Finally, an analysis of the transcryptome will be carried out, which will allow to identify the differential expression of genes and metabolic pathways involved in the immune response and thus to understand how asymptomatic people can control the infection.

ELIGIBILITY:
Inclusion Criteria for asymptomatic careers

* Male and Female
* Age between 18 and 80 years
* PCR and western blot positive to L. Infantum (these exams will be redone as part of the study).
* Signature of informed consent
* Affiliation to a social security scheme

Exclusion Criteria:

* Presence of known immunosuppression or immunosuppressive therapy. -HIV-positive people will be excluded because of the immunosuppressive action of HIV on the immune system. HIV status will be determined by interrogation.
* Pregnant women will be excluded. A urinary pregnancy test (taken from the inclusion proposal) will be performed for women of child-bearing age. The results will be communicated to the patient by a doctor of her choice.
* Persons under guardianship

Inclusion Criteria for healthy patient

* Male or Female
* Age between 18 and 80 years
* PCR and western blot negative Leishmania (these exams will be redone as part of the study).
* Signature of informed consent
* Affiliation to a social security scheme

Exclusion Criteria:

* Presence of known immunosuppression or immunosuppressive therapy. -HIV-positive people will be excluded because of the immunosuppressive action of HIV on the immune system. HIV status will be determined by interrogation.
* Pregnant women will be excluded. A urinary pregnancy test (taken from the inclusion proposal) will be performed for women of child-bearing age. The results will be communicated to the patient by a doctor of her choice.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
immune response of lymphocytes from asymptomatic carriers | 15 months
  decription of immune response of lymphocytes from asymptomatic carriers after stimulation by Leishmania vaccine peptides in ex vivo ELIPSPOT: Presence or absence of immune response.

CONTACTS AND LOCATIONS:
Locations (1):
- Nice Hospital, Nice, France